CLINICAL TRIAL: NCT04816669
Title: A PHASE 3, RANDOMIZED, OBSERVER-BLIND STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF MULTIPLE FORMULATIONS OF THE VACCINE CANDIDATE BNT162B2 AGAINST COVID 19 IN HEALTHY ADULTS 18 THROUGH 55 YEARS OF AGE
Brief Title: A Study to Evaluate Safety, Tolerability, & Immunogenicity of Multiple Formulations of BNT162b2 Against COVID-19 in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C4591020
Record Dates: First submitted 2021-03-24; First posted 2021-03-25 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-11

CONDITIONS: SARS-CoV-2 Infection; COVID-19
Keywords: COVID-19; Coronavirus; Vaccine; SARS-CoV-2; RNA Vaccine
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Lyophilized SDV (Experimental)
  Interventions: Biological: BNT162b2
- Frozen liquid MDV (control for lyo SDV) (Experimental): Control for lyophilized SDV
  Interventions: Biological: BNT162b2
- Frozen-liquid with LNP size at the upper end of specification (Experimental)
  Interventions: Biological: BNT162b2
- RTU (Experimental)
  Interventions: Biological: BNT162b2
- Frozen liquid MDV (given as third dose following a primary series of lyophilized BNT162b2) (Experimental): Additional vaccine dose, using the frozen-liquid formulation, offered to participants who originally received 2 doses of the lyophilized formulation of BNT162b2
  Interventions: Biological: BNT162b2

INTERVENTIONS:
Biological: BNT162b2 — Intramuscular injection

SUMMARY:
This study will compare the safety and tolerability of lyophilized BNT162b2 presented in single dose vials to those of frozen-liquid BNT162b2 in multidose vials and determine whether the immune response is noninferior. Separately, the study will also describe the safety and immunogenicity of frozen-liquid BNT162b2 with lipid nanoparticle size at the upper end of specification and ready to use BNT162b2 (the immediate manufacturing precursor to the lyophilate). Additionally, the study will describe the safety and immunogenicity of an additional dose of frozen liquid BNT162b2 to participants who already received the 2-dose schedule of lyophilized BNT162b2.

* 2-dose schedule (separated by 21 days)
* At a dose of 30µg (as studied in the Phase 2/3 study C4591001)
* In healthy adults 18 through 55 years of age
* The duration of the study for each participant will be approximately 2 months (3 visits in total)
* The study will be conducted in the United States

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants 18 - 55 years of age, inclusive, at Visit 1, (Day 1).
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study. Note: Healthy participants with pre-existing stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 6 weeks before enrolment, can be included.
* Capable of giving personal signed informed consent, which includes compliance with the requirements and restrictions listed in the ICD and in the protocol.
* For Dose 3: Participants who received BOTH doses of the lyophilized formulation of BNT162b2 as part of the initial study.

Exclusion Criteria:

* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Known infection with HIV, HCV, or HBV.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
* Previous clinical (based on COVID-19 symptoms/signs alone, if a SARS-CoV-2 NAAT result was not available) or microbiological (based on COVID-19 symptoms/signs and a positive SARS-CoV-2 NAAT result) diagnosis of COVID-19.
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Women who are pregnant or breastfeeding.
* Previous vaccination with any coronavirus vaccine.
* Receipt of medications intended to prevent COVID-19.
* Individuals who receive treatment with radiotherapy or immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids (if systemic corticosteroids are administered for ≥14 days at a dose of ≥20 mg/day of prednisone or equivalent), eg, for cancer or an autoimmune disease, or planned receipt throughout the study. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
* Receipt of blood/plasma products or immunoglobulin, from 60 days before study intervention administration or planned receipt throughout the study.
* Participation in other studies involving study intervention within 28 days prior to study entry and/or during study participation / Previous participation in other studies involving study intervention containing lipid nanoparticles (LNPs).
* Previous participation in other studies involving study intervention containing lipid nanoparticles.
* Investigator site staff or Pfizer/BioNTech employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 629 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- United States (21):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Research Centers of America ( Hollywood ), Hollywood, Florida
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Solaris Clinical Research, Meridian, Idaho
  - Kentucky Pediatric/ Adult Research, Bardstown, Kentucky
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Amici Clinical Research LLC, Raritan, New Jersey
  - Accellacare (formerly PMG Research of Wilmington, LLC), Wilmington, North Carolina
  - Aventiv Research Inc, Columbus, Ohio
  - Benchmark Research, Austin, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - DM Clinical Research (Administrative and Storage Office only), Tomball, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591020

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted in two parts: Part 1 and Part 2. Participants who received 2 doses of lyophilized formulation of BNT162b2 in Part 1, were offered to receive Dose 3 of frozen-liquid formulation.
Groups:
- BNT162b2 Lyophilized Single Dose Vial (SDV): Part 1: Participants were randomized to receive 30 microgram (mcg) intramuscular dose of lyophilized BNT162b2 in SDV as 2-dose schedule separated by 19 to 23 days. Participants were followed up for safety for 1 month after second dose of vaccine. Participants after receiving 2 doses of lyophilized formulation of BNT162b2 and who consented to receive frozen formulation of BNT162b2, received 30 mcg intramuscular single dose of frozen liquid BNT162b2 in MDV at least 90 days post Vaccination 2. Participants were followed up for safety for 1 month after dose 3.
- BNT162b2 Frozen-Liquid Multi Dose Vial (MDV): Part 1: Participants were randomized to receive 30 mcg intramuscular dose of frozen liquid BNT162b2 in MDV as 2-dose schedule separated by 21 days. Participants were followed up for safety for 1 month after second dose of vaccine.
- BNT162b2 Frozen-Liquid With Lipid Nanoparticle (LNP) Size: Part 2: Participants were randomized to receive 30 mcg intramuscular dose of frozen liquid BNT162b2 with LNP as 2-dose schedule separated by 21 days. Participants were followed up for safety for 1 month after second dose of vaccine.
- BNT162b2 Frozen-Liquid With Ready-to-use (RTU) Size: Part 2: Participants were randomized to receive 30 mcg intramuscular dose of frozen liquid BNT162b2 with RTU as 2-dose schedule separated by 21 days. Participants were followed up for safety for 1 month after second dose of vaccine.
Period: Part 1
Arm/Group | BNT162b2 Lyophilized Single Dose Vial (SDV): Part 1 | BNT162b2 Frozen-Liquid Multi Dose Vial (MDV): Part 1 | BNT162b2 Frozen-Liquid With Lipid Nanoparticle (LNP) Size: Part 2 | BNT162b2 Frozen-Liquid With Ready-to-use (RTU) Size: Part 2
Started | 279 | 280 | 0 | 0
Vaccinated at Dose 1 | 279 | 280 | 0 | 0
Vaccinated at Dose 2 | 276 | 277 | 0 | 0
Vaccination at Dose 3 | 114 (Participants who received 2 doses of lyophilized formulation of BNT162b2 in Part 1, were offered to receive Dose 3 of frozen-liquid formulation.) | 0 | 0 | 0
Completed | 275 | 274 | 0 | 0
Not Completed | 4 | 6 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0
Period: Part 2
Arm/Group | BNT162b2 Lyophilized Single Dose Vial (SDV): Part 1 | BNT162b2 Frozen-Liquid Multi Dose Vial (MDV): Part 1 | BNT162b2 Frozen-Liquid With Lipid Nanoparticle (LNP) Size: Part 2 | BNT162b2 Frozen-Liquid With Ready-to-use (RTU) Size: Part 2
Started | 0 | 0 | 35 | 35
Vaccinated at Dose 1 | 0 | 0 | 35 | 35
Vaccinated at Dose 2 | 0 | 0 | 35 | 35
Completed | 0 | 0 | 33 | 34
Not Completed | 0 | 0 | 2 | 1
Not completed — Other | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population set included all randomized participants who received at least 1 dose of the study intervention.
Groups:
- BNT162b2 Lyophilized SDV: Part 1: Participants were randomized to receive 30 mcg intramuscular dose of lyophilized BNT162b2 in SDV as 2-dose schedule separated by 19 to 23 days. Participants were followed up for safety for 1 month after second dose of vaccine Participants who consented to receive frozen formulation of BNT162b2, received 30 mcg intramuscular single dose of frozen liquid BNT162b2 in MDV at least 90 days post Vaccination 2. Participants were followed up for safety for 1 month after dose 3.
- BNT162b2 Frozen-Liquid MDV: Part 1: Participants were randomized to receive 30 mcg intramuscular dose of frozen liquid BNT162b2 in MDV as 2-dose schedule separated by 21 days. Participants were followed up for safety for 1 month after second dose of vaccine.
- BNT162b2 Frozen-Liquid With LNP Size: Part 2: Participants were randomized to receive 30 mcg intramuscular dose of frozen liquid BNT162b2 with LNP as 2-dose schedule separated by 21 days. Participants were followed up for safety for 1 month after second dose of vaccine.
- BNT162b2 Frozen-Liquid With RTU Size: Part 2: Participants were randomized to receive 30 mcg intramuscular dose of frozen liquid BNT162b2 with RTU as 2-dose schedule separated by 21 days. Participants were followed up for safety for 1 month after second dose of vaccine.
- Total: Total of all reporting groups
Arm/Group | BNT162b2 Lyophilized SDV: Part 1 | BNT162b2 Frozen-Liquid MDV: Part 1 | BNT162b2 Frozen-Liquid With LNP Size: Part 2 | BNT162b2 Frozen-Liquid With RTU Size: Part 2 | Total
Number analyzed (Participants) | 279 | 280 | 35 | 35 | 629
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 279 | 280 | 35 | 35 | 629
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 126 | 20 | 18 | 307
  Male | 136 | 154 | 15 | 17 | 322
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 57 | 55 | 5 | 9 | 126
  Not Hispanic or Latino | 219 | 221 | 30 | 25 | 495
  Unknown or Not Reported | 3 | 4 | 0 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 0 | 2
  Asian | 26 | 16 | 6 | 3 | 51
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 0 | 0 | 5
  Black or African American | 19 | 34 | 2 | 3 | 58
  White | 228 | 220 | 24 | 28 | 500
  More than one race | 3 | 5 | 2 | 0 | 10
  Unknown or Not Reported | 0 | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Full-Length S-Binding IgG Concentrations of Lyophilized Formulation SDVs and Frozen-Liquid Formulation in MDVs 1 Month After Dose 2
Description: GMTs of full-length S-binding IgG level for lyophilized formulation in SDVs and frozen-Liquid formulation in MDVs were reported in this outcome measure as geometric mean concentration (GMCs) in descriptive data section. GMC and 95 percent (%) confidence interval (CI) were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ. Geometric mean ratio (GMR) was calculated as ratios of GMCs of BNT162b2 30 mcg lyophilized SDV and frozen-liquid MDV. GMR are reported in the statistical analysis section.
Time Frame: 1 Month after Dose 2
Population: Evaluable immunogenicity population: Participants who were eligible and randomized, received 2 doses of vaccine, with Dose 2 received within 19 to 42 days after Dose 1, had at least 1 valid immunogenicity result within 28 to 42 days after Dose 2, were negative for both SARS-CoV-2 tests at both Day 1 and 1 month post-Dose 2 visits, and had no other important protocol deviations as determined by clinician.
Measure: Geometric Mean (95% Confidence Interval); unit: Unit per milliliter
Arm/Group | BNT162b2 Lyophilized SDV: Part 1 | BNT162b2 Frozen-Liquid MDV: Part 1
Number analyzed (Participants) | 238 | 226
Unit per milliliter | 4796.8 [4414.1 to 5212.8] | 7031.6 [6393.6 to 7733.3]
Statistical Analysis 1: Comparison: BNT162b2 Lyophilized SDV: Part 1 vs BNT162b2 Frozen-Liquid MDV: Part 1; Test type: Non-Inferiority — Noninferiority was declared if the lower bound of the 2-sided 95% CI for the GMR is greater than 0.67; Geometric mean ratio = 0.68, 95% CI 2-sided [0.60 to 0.77] — GMRs and 2-sided 95% CIs were calculated by exponentiating the mean difference of the logarithms of the concentrations BNT162b2 lyophilized SDV - BNT162b2 frozen-liquid MDV and the corresponding CI (based on the Student t distribution)

2. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 1
Description: Local reactions were collected by the participant using an electronic diary. Local reactions included redness, swelling, and pain at injection site after each vaccination.
Time Frame: Within 7 days after Dose 1
Population: Safety population set included all randomized participants who received at least 1 dose of the study intervention. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BNT162b2 Lyophilized SDV: Part 1 | BNT162b2 Frozen-Liquid MDV: Part 1 | BNT162b2 Frozen-Liquid With Lipid Nanoparticle (LNP) Size: Part 2 | BNT162b2 Frozen-Liquid With Ready-to-use (RTU) Size: Part 2
Number analyzed (Participants) | 278 | 280 | 35 | 35
Percentage of participants
  Redness | 4.0 [2.0 to 7.0] | 5.0 [2.8 to 8.2] | 0 [0.0 to 10.0] | 2.9 [0.1 to 14.9]
  Swelling | 3.6 [1.7 to 6.5] | 3.6 [1.7 to 6.5] | 0 [0.0 to 10.0] | 5.7 [0.7 to 19.2]
  Pain at Injection Site | 78.1 [72.7 to 82.8] | 87.1 [82.6 to 90.8] | 85.7 [69.7 to 95.2] | 68.6 [50.7 to 83.1]

3. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 2
Description: as for outcome 2
Time Frame: Within 7 days after Dose 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BNT162b2 Lyophilized SDV: Part 1 | BNT162b2 Frozen-Liquid MDV: Part 1 | BNT162b2 Frozen-Liquid With Lipid Nanoparticle (LNP) Size: Part 2 | BNT162b2 Frozen-Liquid With Ready-to-use (RTU) Size: Part 2
Number analyzed (Participants) | 274 | 274 | 35 | 35
Percentage of participants
  Redness | 3.6 [1.8 to 6.6] | 5.5 [3.1 to 8.9] | 0 [0.0 to 10.0] | 0 [0.0 to 10.0]
  Swelling | 2.9 [1.3 to 5.7] | 3.3 [1.5 to 6.1] | 0 [0.0 to 10.0] | 8.6 [1.8 to 23.1]
  Pain at Injection Site | 71.2 [65.4 to 76.5] | 80.3 [75.1 to 84.8] | 71.4 [53.7 to 85.4] | 62.9 [44.9 to 78.5]

4. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 1
Description: Systemic events were reported using an electronic diary. Fever was defined as temperature >=38.0 degree Celsius (C). Systemic events including fever, fatigue, headache, chills, new or worsened muscle pain, new or worsened joint pain, vomiting, and diarrhea after Dose 1 were reported.
Time Frame: Within 7 days after Dose 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BNT162b2 Lyophilized SDV: Part 1 | BNT162b2 Frozen-Liquid MDV: Part 1 | BNT162b2 Frozen-Liquid With Lipid Nanoparticle (LNP) Size: Part 2 | BNT162b2 Frozen-Liquid With Ready-to-use (RTU) Size: Part 2
Number analyzed (Participants) | 278 | 280 | 35 | 35
Percentage of participants
  Fever >=38.0 degree C | 0 [0.0 to 1.3] | 3.2 [1.5 to 6.0] | 0 [0.0 to 10.0] | 0 [0.0 to 10.0]
  Fatigue | 46.4 [40.4 to 52.5] | 57.5 [51.5 to 63.4] | 54.3 [36.6 to 71.2] | 45.7 [28.8 to 63.4]
  Headache | 31.3 [25.9 to 37.1] | 44.3 [38.4 to 50.3] | 37.1 [21.5 to 55.1] | 31.4 [16.9 to 49.3]
  Chills | 8.6 [5.6 to 12.6] | 18.6 [14.2 to 23.6] | 8.6 [1.8 to 23.1] | 8.6 [1.8 to 23.1]
  Vomiting | 2.9 [1.3 to 5.6] | 2.1 [0.8 to 4.6] | 5.7 [0.7 to 19.2] | 2.9 [0.1 to 14.9]
  Diarrhea | 14.4 [10.5 to 19.1] | 13.9 [10.1 to 18.5] | 5.7 [0.7 to 19.2] | 11.4 [3.2 to 26.7]
  New or worsened muscle pain | 16.5 [12.4 to 21.4] | 27.1 [22.0 to 32.8] | 11.4 [3.2 to 26.7] | 20.0 [8.4 to 36.9]
  New or worsened joint pain | 7.9 [5.0 to 11.7] | 15.4 [11.3 to 20.1] | 11.4 [3.2 to 26.7] | 17.1 [6.6 to 33.6]

5. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 2
Description: Systemic events were reported using an electronic diary. Fever was defined as temperature >=38.0 degree C. Systemic events including fever, fatigue, headache, chills, new or worsened muscle pain, new or worsened joint pain, vomiting, and diarrhea after Dose 2 were reported.
Time Frame: Within 7 days after Dose 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BNT162b2 Lyophilized SDV: Part 1 | BNT162b2 Frozen-Liquid MDV: Part 1 | BNT162b2 Frozen-Liquid With Lipid Nanoparticle (LNP) Size: Part 2 | BNT162b2 Frozen-Liquid With Ready-to-use (RTU) Size: Part 2
Number analyzed (Participants) | 274 | 274 | 35 | 35
Percentage of participants
  Fever >=38.0 degree C | 6.2 [3.7 to 9.7] | 12.4 [8.7 to 16.9] | 2.9 [0.1 to 14.9] | 5.7 [0.7 to 19.2]
  Fatigue | 60.9 [54.9 to 66.8] | 75.2 [69.6 to 80.2] | 48.6 [31.4 to 66.0] | 60.0 [42.1 to 76.1]
  Headache | 48.2 [42.1 to 54.3] | 61.7 [55.6 to 67.5] | 40.0 [23.9 to 57.9] | 40.0 [23.9 to 57.9]
  Chills | 27.7 [22.5 to 33.4] | 46.4 [40.3 to 52.4] | 22.9 [10.4 to 40.1] | 17.1 [6.6 to 33.6]
  Vomiting | 3.6 [1.8 to 6.6] | 2.2 [0.8 to 4.7] | 2.9 [0.1 to 14.9] | 0 [0.0 to 10.0]
  Diarrhea | 12.8 [9.1 to 17.3] | 14.6 [10.6 to 19.3] | 8.6 [1.8 to 23.1] | 14.3 [4.8 to 30.3]
  New or worsened muscle pain | 32.8 [27.3 to 38.8] | 43.1 [37.1 to 49.2] | 20.0 [8.4 to 36.9] | 37.1 [21.5 to 55.1]
  New or worsened joint pain | 16.8 [12.6 to 21.8] | 32.1 [26.6 to 38.0] | 11.4 [3.2 to 26.7] | 28.6 [14.6 to 46.3]

6. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) From Dose 1 to 1 Month After Dose 2
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect or that was considered to be an important medical event. AEs included all non-SAEs and SAEs. Only AEs collected by non-systematic assessment (i.e. excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: Dose 1 up to 1 Month after Dose 2 (for approximately 2 months)
Population: Safety population set included all randomized participants who received at least 1 dose of the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | BNT162b2 Lyophilized SDV: Part 1 | BNT162b2 Frozen-Liquid MDV: Part 1 | BNT162b2 Frozen-Liquid With Lipid Nanoparticle (LNP) Size: Part 2 | BNT162b2 Frozen-Liquid With Ready-to-use (RTU) Size: Part 2
Number analyzed (Participants) | 279 | 280 | 35 | 35
Participants
  AEs | 16 | 21 | 4 | 4
  SAEs | 0 | 0 | 0 | 0

7. Secondary Outcome: Geometric Mean Concentrations (GMCs) of Full-length S-binding IgG Levels at Baseline: Part 1
Description: GMCs of full-length S-binding IgG levels were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: Baseline (Before Dose 1 on Day 1)
Population: Evaluable immunogenicity population: Participants who were eligible and randomized, received 2 doses of vaccine, with Dose 2 received within 19 to 42 days after Dose 1, had at least 1 valid immunogenicity result within 28 to 42 days after Dose 2, were negative for both SARS-CoV-2 tests at both Day 1 and 1 month post-Dose 2 visits, and had no other important protocol deviations as determined by clinician. "Overall Number of Participants Analyzed": participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Unit per milliliter
Arm/Group | BNT162b2 Lyophilized SDV: Part 1 | BNT162b2 Frozen-Liquid MDV: Part 1
Number analyzed (Participants) | 236 | 226
Unit per milliliter | 2.2 [1.8 to 2.6] | 2.2 [1.8 to 2.6]

8. Secondary Outcome: Geometric Mean Fold Rises (GMFRs) in Full-length S-binding IgG Levels From Baseline to 1 Month After Dose 2: Part 1
Description: GMFRs were defined as ratios of the geometric mean concentration of IgG at 1 month after Dose 2 to the geometric mean concentration of IgG at Baseline. GMFRs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: From Baseline (Before Dose 1 on Day 1) up to 1 Month after Dose 2
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | BNT162b2 Lyophilized SDV: Part 1 | BNT162b2 Frozen-Liquid MDV: Part 1
Number analyzed (Participants) | 236 | 226
Fold rise | 2189.0 [1841.6 to 2601.9] | 3194.0 [2665.8 to 3826.8]

9. Other Pre Specified Outcome: GMTs of Full-Length S-Binding IgG Concentrations of Frozen Liquid With LNP Size at Upper End of Specification and Frozen-Liquid Formulation in MDVs 1 Month After Dose 2
Description: GMTs of full-length S-binding IgG level for frozen liquid with LNP size at upper end of specification relative to frozen-liquid formulation in MDVs were reported in this outcome measure as GMCs in descriptive data section. GMC and 95 % CI were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ. GMR was calculated as ratios of GMCs of BNT162b2 30 mcg frozen liquid with LNP size at upper end of specification relative to frozen-liquid formulation in MDVs. GMR are reported in the statistical analysis section.
Time Frame: 1 Month after Dose 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Unit per milliliter
Arm/Group | BNT162b2 Frozen-Liquid With Lipid Nanoparticle (LNP) Size: Part 2 | BNT162b2 Frozen-Liquid With Ready-to-use (RTU) Size: Part 2
Number analyzed (Participants) | 24 | 28
Unit per milliliter | 7773.3 [5758.5 to 10493.1] | 6839.9 [5242.9 to 8923.5]
Statistical Analysis 1: Comparison: BNT162b2 Frozen-Liquid With Lipid Nanoparticle (LNP) Size: Part 2 vs BNT162b2 Frozen-Liquid With Ready-to-use (RTU) Size: Part 2; Test type: Non-Inferiority — Noninferiority was declared if the lower bound of the 2-sided 95% CI for the GMR is greater than 0.67; Geometric mean ratio = 1.14, 95% CI 2-sided [0.77 to 1.68] — GMRs and 2-sided 95% CIs were calculated by exponentiating the mean difference of the logarithms of the concentrations BNT162b2 frozen-liquid LNP - BNT162b2 frozen-liquid RTU and the corresponding CI (based on the Student t distribution)

10. Other Pre Specified Outcome: GMCs of Full-length S-binding IgG Levels at Baseline and 1 Month After Dose 2: Part 2
Description: as for outcome 7
Time Frame: Baseline (Before Dose 1 on Day 1), 1 Month after Dose 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Unit per milliliter
Arm/Group | BNT162b2 Frozen-Liquid With Lipid Nanoparticle (LNP) Size: Part 2 | BNT162b2 Frozen-Liquid With Ready-to-use (RTU) Size: Part 2
Number analyzed (Participants) | 24 | 28
Unit per milliliter
  Baseline | 2.3 [1.3 to 4.3] | 3.3 [1.6 to 6.7]
  1 Month after Dose 2 | 7773.3 [5758.5 to 10493.1] | 6839.9 [5242.9 to 8923.5]

11. Other Pre Specified Outcome: GMFRs in Full-length S-binding IgG Levels From Baseline to 1 Month After Dose 2: Part 2
Description: as for outcome 8
Time Frame: From Baseline (Before Dose 1 on Day 1) up to 1 Month after Dose 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | BNT162b2 Frozen-Liquid With Lipid Nanoparticle (LNP) Size: Part 2 | BNT162b2 Frozen-Liquid With Ready-to-use (RTU) Size: Part 2
Number analyzed (Participants) | 24 | 28
Fold rise | 3339.1 [1662.6 to 6706.4] | 2072.1 [987.5 to 4348.0]

12. Other Pre Specified Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 3
Description: Local reactions were collected by the participant using an electronic diary. Local reactions included redness, swelling, and pain at injection site after Dose 3.
Time Frame: Within 7 days after Dose 3
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- BNT162b2 Frozen-Liquid MDV: Dose 3: Participants who originally received 2 doses of lyophilized SDV formulation of BNT162b2 30 mcg in Part 1 of the study were administered with an additional dose of frozen liquid MDV of BNT162b2 30 mcg at least 3 months after Dose 2. Participants were followed up for safety for 1 month after third dose of vaccine.
Arm/Group | BNT162b2 Frozen-Liquid MDV: Dose 3
Number analyzed (Participants) | 107
Percentage of participants
  Redness | 6.5 [2.7 to 13.0]
  Swelling | 6.5 [2.7 to 13.0]
  Pain at Injection Site | 70.1 [60.5 to 78.6]

13. Other Pre Specified Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 3
Description: Systemic events were reported using an electronic diary. Fever was defined as temperature >=38.0 degree Celsius (C). Systemic events including fever, fatigue, headache, chills, new or worsened muscle pain, new or worsened joint pain, vomiting, and diarrhea after Dose 3 were reported.
Time Frame: Within 7 days after Dose 3
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BNT162b2 Frozen-Liquid MDV: Dose 3
Number analyzed (Participants) | 107
Percentage of participants
  Fever >=38.0 degree C | 8.4 [3.9 to 15.4]
  Fatigue | 63.6 [53.7 to 72.6]
  Headache | 52.3 [42.5 to 62.1]
  Chills | 39.3 [30.0 to 49.2]
  Vomiting | 2.8 [0.6 to 8.0]
  Diarrhea | 13.1 [7.3 to 21.0]
  New or worsened muscle pain | 29.0 [20.6 to 38.5]
  New or worsened joint pain | 16.8 [10.3 to 25.3]
  Use of antipyretic or pain medication | 35.5 [26.5 to 45.4]

14. Other Pre Specified Outcome: Number of Participants With AEs and SAEs From Dose 3 to 1 Month After Dose 3
Description: as for outcome 6
Time Frame: Dose 3 up to 1 Month after Dose 3 (1 month)
Population: Safety population set included all randomized participants who received at least 1 dose of the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | BNT162b2 Frozen-Liquid MDV: Dose 3
Number analyzed (Participants) | 114
Participants
  AEs | 10
  SAEs | 0

15. Other Pre Specified Outcome: GMFRs in Full-length S-binding IgG Levels From Before Dose 3 to 1 Month After Dose 3
Description: GMFRs were defined as ratios of the geometric mean concentration of IgG from 1 month after Dose 3 to geometric mean concentration of IgG before Dose 3. GMFRs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: From before Dose 3 to 1 Month after Dose 3
Population: Evaluable immunogenicity population:Participants who were eligible and randomized,received 2 doses of lyophilized SDV,with Dose 2 received within 19 to 42 days after Dose 1,received Dose 3 of frozen liquid MDV,had at least 1 valid immunogenicity result within 28 to 42 days after Dose 3,were negative for both SARS-CoV-2 tests at Day 1 and 1 month post-Dose 3 visits, and had no other important protocol deviations as determined by clinician.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | BNT162b2 Frozen-Liquid MDV: Dose 3
Number analyzed (Participants) | 88
Fold rise | 16.0 [13.9 to 18.5]

16. Other Pre Specified Outcome: GMCs of Full-Length S-Binding IgG Levels at Baseline, 1 Month After Dose 2, Before Dose 3, and 1 Month After Dose 3
Description: as for outcome 7
Time Frame: Baseline, 1 Month after Dose 2, before Dose 3, and 1 Month after Dose 3
Population: Evaluable immunogenicity population:Participants eligible and randomized,received 2 doses of lyophilized SDV,with Dose 2 received within 19 to 42 days after Dose 1,received Dose 3 of frozen liquid MDV,had at least 1 valid immunogenicity result within 28 to 42 days after Dose 3,negative for both SARS-CoV-2 tests at Day 1,1 month post Dose 3 visits, had no other important protocol deviations determined by clinician. Here, n= participants evaluable for specific timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Unit per milliliter
Arm/Group | BNT162b2 Frozen-Liquid MDV: Dose 3
Number analyzed (Participants) | 88
Unit per milliliter
  Baseline | 2.1 [1.6 to 2.7]
  1 Month after Dose 2: number analyzed (Participants) | 86
  1 Month after Dose 2 | 4612.2 [4065.7 to 5232.1]
  Before Dose 3 | 874.4 [735.6 to 1039.4]
  1 Month after Dose 3 | 14006.7 [11902.7 to 16482.7]

ADVERSE EVENTS:
Time Frame: AEs and SAEs- For Part 1 and Part 2: Day 1 of Dose 1 up to 1 Month after Dose 2 (approximately2 months); Dose 3: From Dose 3 to 1 Month after Dose 3 (up to 1 month); Local reactions/systemic events (systematic collection): Within 7 days after each dose
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | BNT162b2 Lyophilized SDV: Part 1 | BNT162b2 Frozen-Liquid MDV: Part 1 | BNT162b2 Frozen-Liquid With Lipid Nanoparticle (LNP) Size: Part 2 | BNT162b2 Frozen-Liquid With Ready-to-use (RTU) Size: Part 2 | BNT162b2 Frozen-Liquid MDV: Dose 3
All-Cause Mortality (participants affected / at risk) | 0/279 | 0/280 | 0/35 | 0/35 | 0/114
Serious Adverse Events (participants affected / at risk) | 0/279 | 0/280 | 0/35 | 0/35 | 0/114
Other Adverse Events (participants affected / at risk) | 262/279 | 274/280 | 33/35 | 31/35 | 87/114
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BNT162b2 Lyophilized SDV: Part 1 (N=279) | BNT162b2 Frozen-Liquid MDV: Part 1 (N=280) | BNT162b2 Frozen-Liquid With Lipid Nanoparticle (LNP) Size: Part 2 (N=35) | BNT162b2 Frozen-Liquid With Ready-to-use (RTU) Size: Part 2 (N=35) | BNT162b2 Frozen-Liquid MDV: Dose 3 (N=114)
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Suspected COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 1 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Bacterial vulvovaginitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 64 | 71 | 5 | 7 | 14
Vomiting (VOMITING) (Gastrointestinal disorders) | 16 | 12 | 3 | 1 | 3
Chills (CHILLS) (General disorders) | 84 | 148 | 9 | 9 | 42
Fatigue (FATIGUE) (General disorders) | 199 | 233 | 24 | 24 | 68
Injection site erythema (REDNESS) (General disorders) | 20 | 24 | 0 | 1 | 7
Injection site pain (PAIN) (General disorders) | 240 | 261 | 31 | 28 | 75
Injection site swelling (SWELLING) (General disorders) | 17 | 18 | 0 | 4 | 7
Pyrexia (FEVER) (General disorders) | 17 | 41 | 1 | 2 | 9
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 61 | 103 | 8 | 13 | 18
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 116 | 153 | 9 | 16 | 31
Headache (HEADACHE) (Nervous system disorders) | 162 | 198 | 18 | 19 | 56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BioNTech SE has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/69/NCT04816669/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT04816669/SAP_001.pdf